CLINICAL TRIAL: NCT07132879
Title: Telehealth in MND-Research (TIM-R): A Research Database for MND
Acronym: TIM-R
Status: Recruiting | Type: Observational
Sponsor: University of Sheffield (Other)
Collaborators: LifeArc (Other)
Responsible Party: Sponsor
Other Study IDs: 187038; 340577 (Other: IRAS number)
Record Dates: First submitted 2025-07-09; First posted 2025-08-20 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-06

CONDITIONS: MND (Motor Neurone DIsease)
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 50 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention - Prospective cohort study — No intervention - Prospective cohort study

SUMMARY:
The aim of this study is to implement the Telehealth in MND system as a research database allowing people with MND to take part in research and provide data remotely (TiM-Research).

TiM-Research is an online platform that helps people with MND in the UK take part in research. It brings MND research studies together in one place, making it quick and easy to learn about opportunities to get involved.

What's involved? Participants will receive information about a wide range of research studies that they can sign up for. This could include filling out questionnaires that help researchers understand how MND progresses, providing biosamples (e.g. saliva), or taking part in interviews and focus groups about their experiences. Participants can choose which studies they want to take part in. Participants will also receive updates on research results from the UK MND Research Institute.

Who can take part? People who live with MND and who are based in the UK can sign up for TiM-Research. To join, participants need a computer, phone, or tablet with an internet connection. A family member or carer can help. Participants' information will be kept secure and confidential.

How do participants sign up? Visit the website to find out more or sign up. www.bit.ly/ukmndri-Tim-R.

DETAILED DESCRIPTION:
Background Motor Neuron Disease (MND) is an incurable disease, causing progressive weakness of muscles involving the limbs, speech, and swallowing, leading to progressive disability and eventual respiratory failure. In the UK, there are approximately 5,000 people with MND (pwMND) at any one time. The average life expectancy following diagnosis is two to three years but the course of MND can vary from only a few months to over ten years. The distress and burden of the disease affects pwMND, their family, and carers, and the relentless progression of disability causes social, emotional, and financial strain.

TiM-Care To provide more responsive care for pwMND and their carers, the Telehealth in MND-Care (TiM-C) on MyPathway system was developed. TiM-C is an online system that enables pwMND and their carers to report their symptoms to healthcare professionals (HCPs) from their homes using an app or via the online website. Users are asked to complete symptom questionnaires (e.g., appetite, weight, functional rating, breathing, mental health), answers to which are securely sent to the clinical portal (see figure one).

TiM-C was co-developed with pwMND, carers, and HCPs. The system is easy to use, even for those with significant disabilities, acceptable, and low in burden, taking approximately five minutes per week to complete. 85% of pwMND would recommend TiM to others and 95% would use TiM if they could not travel to clinic. HCPs found it accurate and easy to use.

TiM-Research To provide pwMND greater access to research from the comfort of their own homes, and collect longitudinal data relating to symptoms and treatment, researchers have created Telehealth in MND-Research (TiM-R). TiM-R will send regular symptom questionnaires to pwMND, whilst also enabling invitations to participate in future projects to be sent to those who are eligible. Results from research projects can then be sent back to participants. Anonymised data from the questionnaires will be made available to researchers in a controlled database.

Aim of the project The aim of this project is to create a research database that pwMND can be invited to and submit regular data (i.e., TiM-R). Users can then be invited to research projects and notified of results. Researchers can apply to a Research Management Committee for access to anonymised data.

Project Design PwMND will be invited to TiM-R through two methods. If they are using TiM-C as part of their clinical care, a notification will appear on their account describing the purposes of TiM-R and providing the participant information sheet (PIS). They can then provide consent if they are willing to join TiM-R. If the individual does not want to join TiM-R, they can still use TiM-C to receive clinical care.

If the individual is not using TiM-C as part of their clinical care, they may still join TiM-R by responding to a study advert, which will describe the purposes of the study and a link to the PIS. Advertisements will be distributed through social media, relevant charities (e.g., MND Association), and patient support groups. If willing, the participant can follow links on the PIS to create their TiM-R account, part of which will include providing consent for the purposes of this study.

Regardless of the invitation method, once the participant has consented, they will have access to TiM-R and will start to receive regular research questionnaires (see section 9). They may also receive invitations to other research projects for which they are eligible. For each of these future projects the user can choose whether to participate.

The participant can choose to withdraw from TiM-R at any time without having to give a reason by contacting the Research Management Committee. Contact details will be available through TiM-R. Any withdrawal from TiM-R will not affect participants' ability to use TiM-C.

Researchers can contact the Research Management Committee to gain access to anonymised data collected through TiM-R. The exact process is described in section 12. Providing that the reason for this data usage falls under one of the topics covered by this generic ethical approval (see section 11), researchers will not require their own NHS ethical approval to use this data. If the Research Management Committee agrees access to anonymised data, the researcher will be provided with log in details to a Trusted Research Environment (TRE), where they can perform analyses and write up necessary reports.

Clinical Data collection Once pwMND have created their TiM-R account, they will be asked to complete regular questionnaires. Additional questionnaires may occasionally be added, either by a researcher request or to update the system in line with literature and patient reported outcome measure development. No questionnaire will ask sensitive questions relating to protected characteristics. The addition or removal of a questionnaire will be dependent on a majority decision of the Research Management Committee, who will consider user burden and justification of need for any adaptations.

PwMND who also have a TiM-C account complete regular symptom questionnaires. Researchers will ask these users to consent to the questionnaires to also be uploaded to the research database and used for research purposes, after they have been anonymised. This will be included in the PIS. The questionnaires include the SNAQ, PHQ-8, and GAD-7, however, these may change over the course of this project, depending on the needs of clinical teams using TiM-C.

Research Project Overview The database will support MND researchers inside and outside of the UK and their collaborators. Any outcomes of the research will provide information to improve the care, quality of life, and treatment of pwMND. All academic outputs will be publicly available on a dedicated website.

Only staff and researchers who have completed relevant research data security training will be granted access to TiM-R. The Research Management Committee will be responsible for ensuring that all participant-identifiable data is excluded from available datasets.

ELIGIBILITY:
Inclusion Criteria:

* People living with MND
* Living in the UK

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: People living with MND in the UK
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2024-12-14 (Actual); Primary Completion 2074-12-14 (Estimated); Study Completion 2074-12-14 (Estimated)

PRIMARY OUTCOMES:
ALSFRS-r (Revised Amyotrophic Lateral Sclerosis Functional Rating Scale) | From enrollment, once every 2 months through study completion or participant withdrawal or death (average 2-5 years per participant)
  Functional rating of MND symptoms
  The ALSFRS-R consists of 12 questions, each scored from 0 to 4.
  Minimum Score: The lowest possible score on the scale is 0, representing the worst performance and a total loss of function across all assessed tasks.
  Maximum Score: The highest possible score is 48, which indicates a normal level of function.
  Scoring: A higher score on the scale is a better outcome, as it indicates a greater retention of physical function and a slower progression of the disease. A declining score signifies a worsening of the patient's condition.
Coping Index-ALS | From enrollment, once every 2 months through study completion or participant withdrawal or death (average 2-5 years per participant)
  The Coping Index-ALS (CI-ALS) is a self-report measure used to assess coping abilities in people with amyotrophic lateral sclerosis (ALS).
  The CI-ALS is a 21-item scale that focuses on two key subscales: "coping by self" and "coping with others."
  Minimum and Maximum Values: The scale uses a nomogram to convert raw scores into interval-level measures, but the exact minimum and maximum numerical values of the scale are not consistently reported as a single, simple range like the ALSFRS-R. Instead, the focus is on the subscales and the overall pattern of scores.
  Scoring: A higher score on the CI-ALS generally means a better outcome. A high score indicates a greater use of adaptive, successful coping strategies, which are associated with improved well-being and, in some studies, even longer survival. The scale helps clinicians identify individuals with poor coping mechanisms so they can receive targeted support.
EQ-5D-5L (EuroQol 5-Dimension 5-Level) | From enrollment, once every 2 months through study completion or participant withdrawal or death (average 2-5 years per participant)
  A generic measure of a person's health status. Scale Values and Scoring
  The EQ-5D-5L assesses health across five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension is rated on five levels of severity. The scores can be interpreted in two main ways:
  1. The Descriptive System The descriptive system generates a 5-digit health profile (e.g., 11111 or 55555), where each digit corresponds to one of the five dimensions.
  Minimum Value: A score of 11111 represents the best possible health state, with "no problems" in any dimension.
  Maximum Value: A score of 55555 represents the worst possible health state, with "extreme problems" or being "unable to" in every dimension.
  Scoring: In this system, a lower score (i.e., a smaller number) indicates a better outcome.
D-12 (Dyspnoea-12) | From enrollment, once every 2 months through study completion or participant withdrawal or death (average 2-5 years per participant)
  D-12 is a patient-reported questionnaire designed to measure the severity of breathlessness by assessing both its physical and emotional components.
  The D-12 consists of 12 items, each rated on a 4-point scale: 0 (none), 1 (mild), 2 (moderate), or 3 (severe).
  Minimum Value: The lowest possible score is 0, which indicates no breathlessness in any of the 12 domains.
  Maximum Value: The highest possible score is 36, representing the maximum possible severity of breathlessness.
  Scoring: A higher score on the Dyspnoea-12 indicates a worse outcome, as it signifies a greater severity of breathlessness and its associated physical and emotional impacts.
M-HADS-D (Depression subscale of the Hospital Anxiety and Depression Scale) | From enrollment, once every 2 months through study completion or participant withdrawal or death (average 2-5 years per participant)
  Anxiety and depression
  The M-HADS-D contains seven questions, with each item scored on a 4-point scale ranging from 0 to 3.
  Minimum Value: The lowest possible score is 0, indicating no symptoms of depression.
  Maximum Value: The highest possible score is 21, indicating severe depressive symptoms.
  Scoring: A higher score on the M-HADS-D indicates a worse outcome. The score is interpreted to determine the likelihood and severity of depression, with scores typically categorized as follows:
  0-7: Normal
  8-10: Borderline or possible depression
  11-21: Probable clinical depression
NFI-MND (Neurological Fatigue Index-Motor Neurone Disease) | From enrollment, once every 2 months through study completion or participant withdrawal or death (average 2-5 years per participant)
  Measure of fatigue in people with MND
  The NFI-MND consists of an 8-item summary scale, as well as separate subscales for "energy" and "weakness." Each item is rated on a scale from 0 to 3.
  Minimum Value: The lowest possible score on the 8-item summary scale is 0, indicating no fatigue.
  Maximum Value: The highest possible score on the 8-item summary scale is 24, indicating maximum fatigue.
  Scoring: A higher score on the NFI-MND indicates a worse outcome, as it signifies a greater level of fatigue.
WHOQoLB (World Health Organization Quality of Life-BREF) -Bref stands for 'brief version' | From enrollment, once every 2 months through study completion or participant withdrawal or death (average 2-5 years per participant)
  The WHOQOL-BREF questionnaire is used to calculate four domain scores and two stand-alone items for overall quality of life and general health. Each item is rated on a 5-point scale. The raw scores are then converted to a transformed score for each domain.
  Minimum Value: For the four main domains, the transformed scores range from 4 to 20 or, when scaled to be comparable with other measures, 0 to 100. A score of 0 or 4 represents the worst possible quality of life in that domain.
  Maximum Value: A score of 20 (on the 4-20 scale) or 100 (on the 0-100 scale) represents the best possible quality of life in that domain.
  Scoring: A higher score on the WHOQOL-BREF indicates a better outcome, meaning a higher quality of life. This applies to both the individual domain scores and the scores for overall quality of life and general health.
MND-SWS (Motor Neurone Disease Social Withdrawal Scale) | From enrollment, once every 2 months through study completion or participant withdrawal or death (average 2-5 years per participant)
  Measure of social withdrawal
  Scale Values and Scoring The MND-SWS has two versions: a 10-item version and a 15-item version. Both versions assess the frequency and quality of social interactions.
  Minimum Value: The lowest possible score for the 10-item scale is 0, indicating no social withdrawal. For the 15-item scale, the minimum score is also 0.
  Maximum Value: The highest possible score for the 10-item scale is 40. For the 15-item scale, the maximum score is 60. A higher score indicates a greater degree of social withdrawal.
  Scoring: A higher score on the MND-SWS indicates a worse outcome, as it reflects an increase in social withdrawal and a decrease in social engagement.
RSES (Rosenberg Self-Esteem Scale) | From enrollment, once every 2 months through study completion or participant withdrawal or death (average 2-5 years per participant)
  Self-esteem
  The RSES consists of 10 items, with responses rated on a 4-point Likert scale from "strongly agree" to "strongly disagree."
  Minimum Value: The lowest possible score is 0, indicating the lowest possible self-esteem.
  Maximum Value: The highest possible score is 30, indicating the highest possible self-esteem.
  Scoring: A higher score on the RSES indicates a better outcome, as it reflects a greater level of self-esteem. However, it's worth noting that the scale is often used for descriptive purposes rather than clinical diagnosis, and scores are typically categorized to indicate low, normal, or high self-esteem.
GSE (General Self-efficacy Scale) | From enrollment, once every 2 months through study completion or participant withdrawal or death (average 2-5 years per participant)
  Self-efficacy
  The GSE has 10 items, and each item is rated on a 4-point Likert scale with responses ranging from "not at all true" to "exactly true".
  Minimum Value: The lowest possible score is 10, which indicates a low level of self-efficacy.
  Maximum Value: The highest possible score is 40, which indicates a high level of self-efficacy.
  Scoring: A higher score on the General Self-Efficacy Scale indicates a better outcome, as it signifies a stronger belief in one's ability to cope, persist, and successfully handle challenges.

CONTACTS AND LOCATIONS:
Overall Officials: Chris McDermott, MBChB, FRCP, PhD, Principal Investigator — University of Sheffield
Locations (1):
- University of Sheffield, Sheffield, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Researchers can apply to use anonymised data that TiM-R collects to answer specific research questions. The process of applying for this data is through the UK MND RI Data Catalyst team, full details of which are provided on their website: https://ukmndri.org/

REFERENCES:
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Background] Rolland Y, Perrin A, Gardette V, Filhol N, Vellas B. Screening older people at risk of malnutrition or malnourished using the Simplified Nutritional Appetite Questionnaire (SNAQ): a comparison with the Mini-Nutritional Assessment (MNA) tool. J Am Med Dir Assoc. 2012 Jan;13(1):31-4. doi: 10.1016/j.jamda.2011.05.003. Epub 2011 Jun 23. PMID 21700503
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Hobson E, Baird W, Bradburn M, Cooper C, Mawson S, Quinn A, Shaw PJ, Walsh T, McDermott CJ. Process evaluation and exploration of telehealth in motor neuron disease in a UK specialist centre. BMJ Open. 2019 Oct 22;9(10):e028526. doi: 10.1136/bmjopen-2018-028526. PMID 31640994
- [Background] Whitehead B, O'Brien MR, Jack BA, Mitchell D. Experiences of dying, death and bereavement in motor neurone disease: a qualitative study. Palliat Med. 2012 Jun;26(4):368-78. doi: 10.1177/0269216311410900. Epub 2011 Jun 28. PMID 21712334
- [Background] O'Brien MR, Whitehead B, Jack BA, Mitchell JD. The need for support services for family carers of people with motor neurone disease (MND): views of current and former family caregivers a qualitative study. Disabil Rehabil. 2012;34(3):247-56. doi: 10.3109/09638288.2011.605511. PMID 22087569
- [Background] Hobson EV, Baird WO, Partridge R, Cooper CL, Mawson S, Quinn A, Shaw PJ, Walsh T, Wolstenholme D, Mcdermott CJ. The TiM system: developing a novel telehealth service to improve access to specialist care in motor neurone disease using user-centered design. Amyotroph Lateral Scler Frontotemporal Degener. 2018 Aug;19(5-6):351-361. doi: 10.1080/21678421.2018.1440408. Epub 2018 Feb 16. PMID 29451026
- [Background] Hobson EV, Baird WO, Bradburn M, Cooper C, Mawson S, Quinn A, Shaw PJ, Walsh T, McDermott CJ. Using telehealth in motor neuron disease to increase access to specialist multidisciplinary care: a UK-based pilot and feasibility study. BMJ Open. 2019 Oct 22;9(10):e028525. doi: 10.1136/bmjopen-2018-028525. PMID 31640993
- [Background] Opie-Martin S, Ossher L, Bredin A, Kulka A, Pearce N, Talbot K, Al-Chalabi A. Motor Neuron Disease Register for England, Wales and Northern Ireland-an analysis of incidence in England. Amyotroph Lateral Scler Frontotemporal Degener. 2021 Feb;22(1-2):86-93. doi: 10.1080/21678421.2020.1812661. Epub 2020 Sep 17. PMID 32940088

DOCUMENTS (2):
  • Study Protocol (2024-03-12): https://cdn.clinicaltrials.gov/large-docs/79/NCT07132879/Prot_000.pdf
  • Informed Consent Form (2024-04-30): https://cdn.clinicaltrials.gov/large-docs/79/NCT07132879/ICF_001.pdf